CLINICAL TRIAL: NCT03763396
Title: A Phase 0 Clinical Trial of Two Candidate Azoles (Ketoconazole and Posaconazole) for Patients With Recurrent High Grade Glioma
Brief Title: Azoles Targeting Recurrent High Grade Gliomas
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-5097
Record Dates: First submitted 2018-11-13; First posted 2018-12-04 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Brain Tumor, Recurrent; Cancer, Advanced; Glioma of Brain
Keywords: recurrent high grade glioma, posaconazole, ketoconazole, hexokinase 2 (HK2)
MeSH Terms: conditions — Brain Neoplasms; Neoplasms; Glioma | interventions — Ketoconazole; posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ketoconazole (KCZ) Single Dose Group (Experimental): Single dose 400mg oral tablets 4-24 hours prior to surgery
  Interventions: Drug: Ketoconazole (KCZ)
- Ketoconazole (KCZ) Repeated Dose Group (Experimental): 400mg oral tablets twice a day (BID) for 2-5 days prior to surgery
  Interventions: Drug: Ketoconazole (KCZ)
- Posaconazole (PCZ) Single Dose group (Experimental): Single dose 300 mg delayed release oral tablets 4-24 hours prior to surgery
  Interventions: Drug: Posaconazole (PCZ)
- Posaconazole (PCZ) Repeated Dose group (Experimental): 300 mg delayed release oral tablets twice a day (BID) for day 1; every day thereafter is a single dose of 300 mg delayed release oral tablets. Total treatment time is 7-10 days prior to surgery.
  Interventions: Drug: Posaconazole (PCZ)

INTERVENTIONS:
Drug: Ketoconazole (KCZ) — Oral Tablet
  Arms: Ketoconazole (KCZ) Repeated Dose Group; Ketoconazole (KCZ) Single Dose Group
Drug: Posaconazole (PCZ) — Delayed Release Oral Tablet
  Arms: Posaconazole (PCZ) Repeated Dose group; Posaconazole (PCZ) Single Dose group

SUMMARY:
High-grade gliomas are the most common and aggressive type of brain cancer. Scientists don't fully understand how they grow and spread, and treatments haven't improved much in recent years. However, it's been discovered that these cancers rely heavily on using glucose to maintain their cancerous traits. In lab tests, drugs from the azole class, which target a key step in glucose metabolism, have shown promise in reducing tumor growth in these cancers. Researchers now want to test two of these drugs, ketoconazole and posaconazole, in patients with recurring high-grade gliomas. A small group of these patients will receive either one or several doses of these drugs before undergoing surgery. During the surgery, doctors will measure how much of the drug is present in the brain. They will also study how the drug affects the tumor, particularly its ability to process glucose. This research aims to provide initial insights into how these drugs work in patients with this type of brain cancer, which could guide future research and treatment strategies.

DETAILED DESCRIPTION:
High grade gliomas (WHO grade III and IV)(HGG) are the most common malignant, and aggressive brain tumour in humans. Current understanding of the mechanisms contributing to their growth and progression remain limited. Furthermore, treatment options have not advanced in recent decades. Recently, it has become evident that these tumours are dependent on glucose metabolism to maintain oncogenic properties. From a preclinical standpoint, targeting hexokinase 2 (HK2), the first committed step of glucose metabolism, with azole class drugs has been shown to display favourable anti-tumour effects in both in vitro and in vivo HGG models. We would like to translate these preclinical findings into the clinical setting by implementing a proof-of biological concept study with two azole drugs: ketoconazole (KCZ) and posaconazole (PCZ). A small cohort of recurrent HGG patients will receive either a single-, or repeated, steady state dose of either KCZ or PCZ and will then go for surgery where drug concentrations will be measured intraoperatively. Study drug selection and dosing details will be selected based on urgency of surgery and patient clinical characteristics Downstream biological effects of drug on tumour tissue, including HK2 activity, will also be assessed. This study will provide a preliminary understanding of azole drug activity in recurrent HGG patients and will help inform future studies of azole drug efficacy in this patient population

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Evidence of recurrent HGG that in the opinion of the treating team does not represent pseudoprogression and would require surgical resection
* Karnofsky Performance Score (KPS) ≥ 60%
* ECOG ≤ 2
* Life expectancy greater than 12 weeks
* Adequate liver function defined as ALT, AST, ALP, GGT, bilirubin within 1.5x institutional upper limit of normal
* Potassium, calcium, and magnesium within normal limits (PCZ cohort)
* Adequate renal function defined as eGFR levels within 1.5x the institutional upper limit of normal (only for KCZ cohort)
* Ability to swallow medication
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation.
* Ability to understand and willingness to sign a written informed consent document
* Be able to comply with treatment plan, study procedures and follow-up examinations

Exclusion Criteria:

* 1. Patients may not be receiving any other investigational agents while on study
* Patients who have known allergy to KCZ, PCZ, or other azoles
* Patients who have previously had a severe side effect, such as agranulocytosis and neutropenia, in conjunction with previous azole class drugs for a parasitic infection
* Patients with a history of acute or chronic hepatitis
* Patients with liver enzymes (ALT, AST, ALP, GGT, Bilirubin) >1.5x above normal range for the laboratory performing the test
* ECG with QT > 450 msec (PCZ cohort)
* Patients taking drugs known to prolong the QT interval (PCZ cohort)
* Patients who are taking metronidazole and cannot be safely moved to a different antibiotic greater than 7 days prior to starting KCZ therapy
* Patients who have taken any azoles within the last 3 months
* Patients who are taking any anti-convulsant medication that interferes with the cytochrome P450 pathway (e.g. phenytoin, phenobarbital, carbamazepine, etc.) and who cannot be switched to alternative medications such as keppra (levetiracetam)
* Uncontrolled intercurrent illness such as chronic hepatitis, acute hepatitis, or psychiatric illness/social situation that would limit compliance with study requirements
* Patients with a history of Addison's disease or other forms of adrenal insufficiency
* Patient with little or no stomach acid production (achlorhydria) are excluded from the KCZ cohort
* Pregnant and breast feeding women
* Patients with a history of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with the study participation or investigational product administration or may interfere with the interpretation of the results.
* Patients who are not available for follow-up assessments or unable to comply with study requirements.
* Patients who are currently taking medications that induce the metabolism of KCZ or PCZ, such as isoniazid, nevirapine, rifamycins (such as rifabutin, rifampin), St. John's wort, among others (see section 5.3 for full details).
* Patients who are currently taking medications for which the metabolism may be affected by KCZ or PCZ, which include but are not limited to: benzodiazepines (such as alprazolam, midazolam, triazolam), domperidone, eletriptan, eplerenone, ergot drugs (such as ergotamine), nisoldipine, drugs used to treat erectile dysfunction-ED or pulmonary hypertension (such as sildenafil, tadalafil), some drugs used to treat seizures (such as carbamazepine, phenytoin), some statin drugs (such as atorvastatin, lovastatin, simvastatin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Intratumoral concentrations of KCZ or PCZ | Following either single dose regimen(4-24hours prior to surgery) or repeated dose regimen of KCZ( for 2-5 days) or PCZ( for 7-10 days)
Plasma concentrations of KCZ or PCZ | Following either single dose regimen(4-24hours prior to surgery) or repeated dose regimen of KCZ(for 2-5 days) or PCZ(for 7-10 days)

SECONDARY OUTCOMES:
Assess Hexokinase 2 activity | Following either single dose regimen(4-24hours prior to surgery) or repeated dose regimen of KCZ(for 2-5 days) or PCZ(for 7-10 days) compared to archive tumor tissue from baseline
  enzyme activity measured using optical absorbance with a spectrophotometer
Assess the biological effects of KCZ or PCZ on metabolites within the glycolytic pathway | Following either single dose regimen(4-24hours prior to surgery) or repeated dose regimen of KCZ(for 2-5 days) or PCZ(for 7-10 days) compared to archive tumor tissue from baseline
  quantify presence/absence of metabolites using mass spectrometry
assess the biological effects of KCZ or PCZ on tumor proliferation | Following either single dose regimen(4-24hours prior to surgery) or repeated dose regimen of KCZ(for 2-5 days) or PCZ(for 7-10 days) compared to archive tumor tissue from baseline
  measured using ki-67 proliferation index
assess biological effects of KCZ or PCZ on tumor cell death | Following either single dose regimen(4-24hours prior to surgery) or repeated dose regimen of KCZ(for 2-5 days) or PCZ(for 7-10 days) compared to archive tumor tissue from baseline
  measured using TUNEL staining
assess biological effects of KCZ or PCZ on tumor angiogenesis | Following either single dose regimen(4-24hours prior to surgery) or repeated dose regimen of KCZ(for 2-5 days) or PCZ(for 7-10 days) compared to archive tumor tissue from baseline
  measured using VEGF/CD-31 immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Gelareh Zadeh, MD, PhD, Principal Investigator — University Health Network/Toronto Western Hospital
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No